CLINICAL TRIAL: NCT05430256
Title: The Early Life Clinical Feature and Risk Factors Analysis Using Artificial Intelligence in Children With Neurodevelopmental Disorders: Premature Infants Cohort Study
Brief Title: The Early Life Clinical Feature and Risk Factors Analysis in Children With Neurodevelopmental Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201801537A3
Record Dates: First submitted 2022-05-30; First posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-04

CONDITIONS: Premature Infant
Keywords: Attention Deficit Hyperactivity Disorder; Autism Spectrum Disorder; Artificial intelligence
MeSH Terms: conditions — Premature Birth; Attention Deficit Disorder with Hyperactivity; Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Premature children with neurological developmental disorder(such as ADHD): Premature children with neurological developmental disorder (such as ADHD): n = 200
- Premature children with neurological developmental disorder(such as ASD): Premature children with neurological developmental disorder (such as ASD): n = 50
- Premature infants with no neurodevelopmental disorders: Premature infants with no neurodevelopmental disorders: n = 200
- Age and gender match in non-preterm children: Age and gender match in non-preterm children: n = 200

SUMMARY:
The study will be a 5-year retrospective and prospective case control study, included 650 participants, and participants will be divided into four groups.By this research the investigators will achieve several aims:(1) Through the cross-sectional analysis of this study, the investigators can understand the current prevalence of developmental disorders in Taiwan ,especially ADHD and ASD, and the ratio of male to female in school-age children. (2) Analysis of risk factors in preterm infants during pregnancy and infant, and construct the diagnostic predictive models. (3) By the cohort study of premature infants, to analyze early risk factors of premature children with neurological developmental disorders (such as ADHD), and develop the diagnostic predictive models and early interventional tools. (4) Using artificial intelligence and machine learning analysis to analyze the characteristics of preterm and development of diagnostic prediction model of premature infant or premature children combined ADHD. (5) The application of noninvasive physiological signal capture real-time analysis system in screening and evaluation of "premature infant and neurodevelopmental disorders".

DETAILED DESCRIPTION:
In recent years the issue of low birth rates become more and more serious in many countries. In 2017, the average birth rate is 1.17 for every child-bearing woman in Taiwan, ranking the last among Asian countries. As the declining birth rates, the population of Taiwan will decrease year by year while showing an aging society. It will be an important crisis in Taiwan's future development. Although the declining birth rates in Taiwan year by year, the incidence of premature has not decrease. Moreover, the morbidity and long-term prognosis of preterm infants, will be a significant burden of children, families, and national economy. Therefore, it should be a serious issue of government. According to the above reasons, to keep the "safe pregnancy and normal development of the fetus," "smooth delivery" and even "postpartum newborn healthy growth" and so on, will be very important issues in the future.

Due to advances in medical technology and the improvement of newborn care, makes the very low birth weight preterm infant survival rate greatly improved. However, the improvement of survival rate did not improve the incidence of postnatal morbidity of the preterm infants, and the risk of many neurodevelopmental disorders greatly increased. Many studies have confirmed the long-term prognosis of preterm infants with low birth weight, whom with serious abnormalities in neurocognitive development, language development, motor development and so on. Attention deficit hyperactivity disorder (ADHD) and Autism spectrum disorder (ASD) are common neurodevelopmental disorders. These deficiencies such as inattention, decreased learning ability, behavioral problems and social skills disturbance ....make the children have poor outcome. It is affect children academic achievement and adaptation so great in the future. Therefore, the government, experts and scholars should concern about the issue of the premature and these pediatric neurological development delay and poor prognosis.

Meanwhile, this study will design a 5-year retrospective and prospective case control study, will include 650 participant. And participants will be divided into four groups:(a) Premature children with neurological developmental disorder (such as ADHD): n = 200; (b) Premature children with neurological developmental disorder (such as ASD): n = 50; (c) Premature infants with no neurodevelopmental disorders: n = 200; (d) Age and gender match in non-preterm children: n = 200.

By this research to achieve the aims: (1) Through the cross-sectional analysis of this study, the investigators can understand the current prevalence of developmental disorders in Taiwan ,especially ADHD and ASD, and the ratio of male to female in school-age children. (2) Analysis of risk factors in preterm infants during pregnancy and infant, and construct the diagnostic predictive models. (3) By the cohort study of premature infants, to analyze early risk factors of premature children with neurological developmental disorders (such as ADHD), and develop the diagnostic predictive models and early interventional tools. (4) Using artificial intelligence and machine learning analysis to analyze the characteristics of preterm and development of diagnostic prediction model of premature infant or premature children combined ADHD. (5) The application of noninvasive physiological signal capture real-time analysis system in screening and evaluation of "premature infant and neurodevelopmental disorders".

ELIGIBILITY:
Inclusion Criteria:

1. The investigators will collect newborns who born in Chang Gung after 2010 .
2. The investigators will collect 450 premature infants under 37 weeks and 200 non-preterm infants.
3. Participated in the former Ministry of Science and Technology research project ''NSC 101-2314-B-182A-072-MY3'' and project ''106-2314-B-182A-040-MY3'' will be invited to join this study.
4. Parents are willing to sign the subject's consent form.

Exclusion Criteria:

1. If children have serious neurological diseases, serious heart problems or serious mental retardation, they will not be able to participate in this study.
2. If parents cannot sign the consent form of the subjects.

Ages: 1 Year to 15 Years | Sex: All
Age Groups: Child
Study Population: 450 premature infants under 37 weeks and 200 non-preterm infants.
Sampling Method: Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2019-04-29 (Actual); Primary Completion 2022-10-16 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Polysomnography (PSG) | Once a year until the study is completed(up to 3 years)
  Change in sleep status based on PSG during the study.
Wechsler Intlligence Scale for Children (WISC) | Once a year until the study is completed(up to 3 years)
  Change in speech comprehension, perceptual reasoning, working memory, and processing speed abilities based on WISC during the study.
  * This assessment will provide a composite score that represents a child's overall intellectual ability (FSIQ),with higher scores indicating better intellectual ability .

SECONDARY OUTCOMES:
OSA-18 questionnaire (OSA-18) | Twice a year until the study is completed(up to 3 years)
  The OSA-18 is a caregiver-administered quality of life survey that contains 18 items divided into five subscales: sleep disturbance, physical symptoms, emotional distress, daytime function, and caregiver concerns. Each item is scored on a seven-point ordinal scale.The OSA-18 total score is the sum of the 18 items, and therefore ranges from 18 (no impact on quality of life) to 126 (major negative impact).
Children's Sleep Habits Questionnaire (CSHQ) | Twice a year until the study is completed(up to 3 years)
  The CSHQ is a parent-rated questionnaire comprised of 45 items; 33 scored questions, and 7 additional items intended to provide other relevant information pertaining to sleep behavior, each scored question is rated on a 3-point scale .Ratings are combined to form eight subscales: Bedtime Resistance, Sleep Onset Delay, Sleep Duration, Sleep Anxiety, Night Wakings, Parasomnias, Sleep Disordered Breathing, and Daytime Sleepiness.With higher scores indicating more sleep problems .
Disruptive Behaviour Disorder Rating Scale (DBDRS) | Twice a year until the study is completed(up to 3 years)
  The DBD parent/teacher rating scale is a screening tool designed to aid in the diagnostic process for a number of child psychopathologies, particularly externalising disorders.The DBD rating scale consists of 42 items related to symptoms of Conduct disorder (16 items), ODD (8 items), ADHD-Inattention (9 items), ADHD- hyperactivity/ Impulsivity (9 items).Each item is rated on a four-point scale ranging from not at all (0) to very much (3).The higher score the child gets, the more behavioral problems he/she has.
Conners' Continuous Performance Test (CPT) | Twice a year until the study is completed(up to 3 years)
  The Conners Continuous Performance Test is a computer administered test that is designed to assess problems with attention.Many statistics are computed including omission errors , commission errors, hit reaction time, hit reaction time standard error, detectability, response style, perseverations , hit reaction time by block, standard error by block, reaction time by ISI , and standard error by ISI. These statistics are converted to T-scores and can be interpreted in terms of various aspects of attention including inattention, impulsivity, and vigilance.Higher rates of correct detections indicate better attentional capacity.
Wisconsin Card Sorting Test (WCST) | Twice a year until the study is completed(up to 3 years)
  The Wisconsin Card Sorting Test (WCST) is a neuropsychological test that is frequently used to measure such higher-level cognitive processes as attention, perseverance,working memory, abstract thinking and set shifting.
Actigraphy | baseline
  Understand the patient's activity and sleep status.
Allergen Test | baseline
  The investigaters plan to draw about 5-10 milliliters of blood for individual subjects to analyze total immunoglobulin E and specific immunoglobulin E for 40 common allergens in the environment.
Di(2-ethylhexyl)phthalate test (DEHP) | baseline
  This project is expected to use the remaining serum and urine of allergens in individual cases, and use the QTRAP® 5500 mass spectrometer system (AB SCIEX) to analyze the concentrations of common plasticizer metabolites.
Child Behavior Checklist (CBCL) | Twice a year until the study is completed(up to 3 years)
  The Child Behavior Checklist (CBCL) is a widely used questionnaire to assess behavioral and emotional problems.The CBCL's questions are associated with problems on a syndrome scale in eight different categories: anxious/depressed, withdrawn/depressed, somatic complaints, social problems, thought problems, attention problems, rule-breaking behavior, and aggressive behavior.According to the normative data of the CBCL, a t-score ≤ 59 indicates non-clinical symptoms, a t-score between 60 and 64 indicates that the child is at risk for problem behaviors, and a t-score ≥ 65 indicates clinical symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Shu Huang, PhD, Study Director — Principal Investigator
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Accornero VH, Amado AJ, Morrow CE, Xue L, Anthony JC, Bandstra ES. Impact of prenatal cocaine exposure on attention and response inhibition as assessed by continuous performance tests. J Dev Behav Pediatr. 2007 Jun;28(3):195-205. doi: 10.1097/01.DBP.0000268560.72580.f9. PMID 17565286
- [Result] Adde L, Helbostad JL, Jensenius AR, Taraldsen G, Grunewaldt KH, Stoen R. Early prediction of cerebral palsy by computer-based video analysis of general movements: a feasibility study. Dev Med Child Neurol. 2010 Aug;52(8):773-8. doi: 10.1111/j.1469-8749.2010.03629.x. Epub 2010 Feb 24. PMID 20187882
- [Result] Batton DG, DeWitte DB, Pryce CJ. One hundred consecutive infants born at 23 weeks and resuscitated. Am J Perinatol. 2011 Apr;28(4):299-304. doi: 10.1055/s-0030-1268714. Epub 2010 Nov 29. PMID 21117014
- [Result] Biederman J, Monuteaux MC, Mick E, Spencer T, Wilens TE, Silva JM, Snyder LE, Faraone SV. Young adult outcome of attention deficit hyperactivity disorder: a controlled 10-year follow-up study. Psychol Med. 2006 Feb;36(2):167-79. doi: 10.1017/S0033291705006410. PMID 16420713
- [Result] Brisson J, Martel K, Serres J, Sirois S, Adrien JL. Acoustic analysis of oral productions of infants later diagnosed with autism and their mother. Infant Ment Health J. 2014 May-Jun;35(3):285-95. doi: 10.1002/imhj.21442. Epub 2014 Mar 31. PMID 25798482
- [Result] Bohm HV, Stewart MG, Healy AM. On the Autistic Spectrum Disorder concordance rates of twins and non-twin siblings. Med Hypotheses. 2013 Nov;81(5):789-91. doi: 10.1016/j.mehy.2013.08.019. Epub 2013 Aug 29. PMID 24055096
- [Result] Canela C, Buadze A, Dube A, Eich D, Liebrenz M. Skills and compensation strategies in adult ADHD - A qualitative study. PLoS One. 2017 Sep 27;12(9):e0184964. doi: 10.1371/journal.pone.0184964. eCollection 2017. PMID 28953946
- [Result] Chu SM, Tsai MH, Hwang FM, Hsu JF, Huang HR, Huang YS. The relationship between attention deficit hyperactivity disorder and premature infants in Taiwanese: a case control study. BMC Psychiatry. 2012 Jul 23;12:85. doi: 10.1186/1471-244X-12-85. PMID 22824325
- [Result] Colvert E, Tick B, McEwen F, Stewart C, Curran SR, Woodhouse E, Gillan N, Hallett V, Lietz S, Garnett T, Ronald A, Plomin R, Rijsdijk F, Happe F, Bolton P. Heritability of Autism Spectrum Disorder in a UK Population-Based Twin Sample. JAMA Psychiatry. 2015 May;72(5):415-23. doi: 10.1001/jamapsychiatry.2014.3028. PMID 25738232
- [Result] DiMaio S, Grizenko N, Joober R. Dopamine genes and attention-deficit hyperactivity disorder: a review. J Psychiatry Neurosci. 2003 Jan;28(1):27-38. PMID 12587848
- [Result] DeVilbiss EA, Gardner RM, Newschaffer CJ, Lee BK. Maternal folate status as a risk factor for autism spectrum disorders: a review of existing evidence. Br J Nutr. 2015 Sep 14;114(5):663-72. doi: 10.1017/S0007114515002470. Epub 2015 Aug 5. PMID 26243379
- [Result] Faustman EM, Silbernagel SM, Fenske RA, Burbacher TM, Ponce RA. Mechanisms underlying Children's susceptibility to environmental toxicants. Environ Health Perspect. 2000 Mar;108 Suppl 1(Suppl 1):13-21. doi: 10.1289/ehp.00108s113. PMID 10698720
- [Result] Fischl B, Dale AM. Measuring the thickness of the human cerebral cortex from magnetic resonance images. Proc Natl Acad Sci U S A. 2000 Sep 26;97(20):11050-5. doi: 10.1073/pnas.200033797. PMID 10984517
- [Result] Ghiassian S, Greiner R, Jin P, Brown MR. Using Functional or Structural Magnetic Resonance Images and Personal Characteristic Data to Identify ADHD and Autism. PLoS One. 2016 Dec 28;11(12):e0166934. doi: 10.1371/journal.pone.0166934. eCollection 2016. PMID 28030565
- [Result] Hallmayer J, Cleveland S, Torres A, Phillips J, Cohen B, Torigoe T, Miller J, Fedele A, Collins J, Smith K, Lotspeich L, Croen LA, Ozonoff S, Lajonchere C, Grether JK, Risch N. Genetic heritability and shared environmental factors among twin pairs with autism. Arch Gen Psychiatry. 2011 Nov;68(11):1095-102. doi: 10.1001/archgenpsychiatry.2011.76. Epub 2011 Jul 4. PMID 21727249
- [Result] Iannaccone R, Hauser TU, Ball J, Brandeis D, Walitza S, Brem S. Classifying adolescent attention-deficit/hyperactivity disorder (ADHD) based on functional and structural imaging. Eur Child Adolesc Psychiatry. 2015 Oct;24(10):1279-89. doi: 10.1007/s00787-015-0678-4. Epub 2015 Jan 23. PMID 25613588
- [Result] Kato I, Groswasser J, Franco P, Scaillet S, Kelmanson I, Togari H, Kahn A. Developmental characteristics of apnea in infants who succumb to sudden infant death syndrome. Am J Respir Crit Care Med. 2001 Oct 15;164(8 Pt 1):1464-9. doi: 10.1164/ajrccm.164.8.2009001. PMID 11704597
- [Result] Mazaheri A, Fassbender C, Coffey-Corina S, Hartanto TA, Schweitzer JB, Mangun GR. Differential oscillatory electroencephalogram between attention-deficit/hyperactivity disorder subtypes and typically developing adolescents. Biol Psychiatry. 2014 Sep 1;76(5):422-9. doi: 10.1016/j.biopsych.2013.08.023. Epub 2013 Oct 8. PMID 24120092
- [Result] Larroque B, Ancel PY, Marret S, Marchand L, Andre M, Arnaud C, Pierrat V, Roze JC, Messer J, Thiriez G, Burguet A, Picaud JC, Breart G, Kaminski M; EPIPAGE Study group. Neurodevelopmental disabilities and special care of 5-year-old children born before 33 weeks of gestation (the EPIPAGE study): a longitudinal cohort study. Lancet. 2008 Mar 8;371(9615):813-20. doi: 10.1016/S0140-6736(08)60380-3. PMID 18328928